CLINICAL TRIAL: NCT01452698
Title: A Phase 3, Randomized, Double-Blind, Multicenter Study to Evaluate the Efficacy and Safety of TAK-438 (20 mg Once-Daily) Compared to AG-1749 (30mg Once-Daily) in Patients With Erosive Esophagitis
Brief Title: Efficacy of TAK-438 Compared to AG-1749 (Lansoprazole) in the Treatment of Erosive Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-438/CCT-002; U1111-1123-8356 (Registry Identifier: WHO); JapicCTI-111607 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2011-09-16; First posted 2011-10-17 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Erosive Esophagitis
Keywords: Drug Therapy
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAK-438 20 mg QD (Experimental)
  Interventions: Drug: TAK-438; Drug: Placebo
- AG-1749 30 mg QD (Active Comparator)
  Interventions: Drug: Lansoprazole; Drug: Placebo

INTERVENTIONS:
Drug: TAK-438 — TAK-438 20 mg, tablets, orally, once daily for up to 8 weeks.
  Arms: TAK-438 20 mg QD
Drug: Placebo — Lansoprazole placebo-matching capsules, orally, once daily for up to 8 weeks.
  For participants whose EE is not endoscopically healed at Week 8, the participants will receive additional treatment of TAK-438 40 mg, tablets, orally, once daily for up to an additional 8 weeks.
  Other Names: AG-1749
  Arms: TAK-438 20 mg QD
Drug: Lansoprazole — Lansoprazole 30 mg, capsules, orally, once daily for up to 8 weeks.
  For participants whose EE is not endoscopically healed at Week 8, the participants will receive additional treatment of TAK-438 40 mg, tablets, orally, once daily for up to an additional 8 weeks.
  Other Names: AG-1749
  Arms: AG-1749 30 mg QD
Drug: Placebo — TAK-438 placebo-matching tablets, orally, once daily for up to 8 weeks.
  Arms: AG-1749 30 mg QD

SUMMARY:
The purpose of this study is to determine the efficacy of TAK-438, once daily (QD), compared to lansoprazole in patients with erosive esophagitis of Grade A to D as defined by the LA classification grading system.

ELIGIBILITY:
Inclusion Criteria:

1. At Visit 1 (start of the observation period), the participant must have endoscopically confirmed erosive esophagitis of Grade A to D, as defined by the LA classification grading system, and the target number of participants who are clearly Grade C or D is 30% (120 participants) or more of the total participants.
2. Outpatient (including inpatient for examination)

Exclusion Criteria:

1. Participants with an esophagus-related complication (eosinophilic esophagitis, esophageal varices, scleroderma, viral or fungal infection, esophageal stenosis, etc.), a history of radiotherapy or cryotherapy of the esophagus, a caustic or physiochemical trauma (esophageal sclerotherapy, etc.). However, participants with Schatzki's ring (mucosal tissue ring around inferior esophageal sphincter) or Barrett's esophagus are allowed to be included.
2. Participants who have received surgery or treatment affecting gastroesophageal reflux (cardioplasty, dilation of esophageal stenosis [excluding Schatzki's ring], etc.), or who have a history of surgery of stomach or duodenum (excluding removal of benign polyp under endoscopy)
3. Participants who have acute upper gastrointestinal bleeding, gastric or duodenal ulcer (mucosal defect with white coating) within 30 days prior to Visit 1 (start of the observation period). However, participants with gastric or duodenal erosions are allowed to be included.
4. Participants with a previous or current history of Zollinger-Ellison syndrome, or other gastric acid hypersecretion disorders

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Endoscopic Healing Rate Over 8 Weeks of Erosive Esophagitis | 8 Weeks
  Endoscopic healing of erosive esophagitis is defined as those participants who have endoscopically confirmed EE of Grade O as defined by the Los Angeles (LA) Classification Grading System. The definitions of each grade are: Grade O (No mucosal break), Grade A (Mucosal break <5 mm), Grade B (Mucosal break ≥5 mm), Grade C (Mucosal break continuous between two or more folds and <75% of the circumference) and Grade D (Mucosal break ≥75% of the circumference).

SECONDARY OUTCOMES:
Endoscopic Healing Rate Over 2 Weeks of Erosive Esophagitis | 2 Weeks
Endoscopic Healing Rate Over 4 Weeks of Erosive Esophagitis | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Senior Manager, Study Director — Takeda
Locations (32):
- Japan (32):
  - Nagoya, Aichi-ken
  - Abiko-shi, Chiba
  - Fukuoka, Fukuoka
  - Itoshima-shi, Fukuoka
  - Kurume-shi, Fukuoka
  - Onga-gun, Fukuoka
  - Gifu, Gifu
  - Annaka-shi, Gunma
  - Aki-gun, Hiroshima
  - Hiroshima, Hiroshima
  - Sapporo, Hokkaido
  - Amagasaki-shi, Hyōgo
  - Kobe, Hyōgo
  - Takarazuka-shi, Hyōgo
  - Sakade-shi, Kagawa-ken
  - Yokohama, Kanagawa
  - Kochi, Kochi
  - Susaki-shi, Kochi
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Nagasaki, Nagasaki
  - Ōita, Oita Prefecture
  - Okayama, Okayama-ken
  - Fuziidera-shi, Osaka
  - Shizuoka, Shizuoka
  - Otawara-shi, Tochigi
  - Chiyoda-ku, Tokyo
  - Chuo-ku, Tokyo
  - Nakano-ku, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Yamagata, Yamagata